CLINICAL TRIAL: NCT07036094
Title: Relationship Between Nutritional Consumption of Breastfeeding Mothers and Breast Milk Composition During Lactation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Breast Milk Composition
Record Dates: First submitted 2025-05-22; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Breastmilk; Breastmilk Expression; Maternal Nutrition
Keywords: human milk; maternal nutrition; lactation; breastmilk
MeSH Terms: conditions — Breast Milk Expression; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hand expressing breast milk (Experimental): Manual milking: Milk was expressed by hand until the milk flow stopped at the mother's breast. While the baby was suckling from one breast, milking was done from the other breast, and a 10 cc sample was taken from the collected milk and placed in sterile fallopian tubes.
  Interventions: Other: Manual breast milk expression

INTERVENTIONS:
Other: Manual breast milk expression — Manual breast milk expression: Milk was expressed by hand until the milk flow stopped at the mother's breast. While the baby was suckling from one breast, milk was expressed from the other breast, and a 10 cc sample was taken from the collected milk and placed in sterile fallopian tubes.
  The mothers' food records were analyzed for 3 days before the milk sample was taken and on the day the milk sample was taken.

SUMMARY:
This study seeks to answer the question of the effect of maternal diet during lactation on breast milk composition. This study was conducted with 31 mothers who were hospitalized in Şanlıurfa Education and Research Hospital due to childbirth between 2024-2025. A nutrition plan was applied to the mothers three days before milk samples were taken and on milking days. Milk was milked by hand milking. Data were obtained with the Introductory Information Form, Breast Milk Information Form, Breast Milk Follow-up Form and Daily Food Consumption Record Form. Frozen milk samples were analyzed with Miris® HMATM to determine protein, fat, carbohydrate and energy values. Data were analyzed using the R programming language version 4.4.1.

DETAILED DESCRIPTION:
Breast milk is the best source of nutrition for infants because it contains essential nutrients and other bioactive factors (e.g., hormones, antibodies, bioactive molecules, stem cells) in the right balance. The macronutrient values in breast milk of mature term babies have been reported as protein 0.9-1.2 gr/dl, fat 3.2-3.6 gr/dl, lactose 6.7-7.8 gr/dl. . It is known that exclusive breastfeeding in the first six months of life and breastfeeding with complementary foods at two years of age and beyond is associated with a reduced incidence of infections and chronic diseases . Studies have shown that breastfeeding has short- and long-term benefits and protective effects. It is known that breast milk protects the baby from chronic diseases, especially Type 1 and Type 2 diabetes, obesity, hypertension, cardiovascular diseases, hyperlipidemia and some types of cancer , has positive effects on the cognitive development of the baby , and this effect continues for many years. These protective effects are controversial and may differ according to maternal phenotypes . Compared to infant formulas with standardized compositions, the composition of breast milk changes dynamically because it is produced by women with significantly different genotypes and phenotypes . The composition of breast milk is affected by many maternal, infant and physiological factors. Some of these factors vary according to whether the baby is term or preterm, whether the milk is colostrum secreted in the first 5 days after birth, transitional milk secreted between 5 days and 2 weeks, and mature milk produced after the 2nd week, the mother's nutritional status, body mass index, parity, gender of the baby, birth weight of the baby, duration of breastfeeding, and the method of milk delivery (expressing/breastfeeding), etc.. However, the effect of maternal nutrition on breast milk composition has not been well defined. There are some limitations in previous studies evaluating the relationship between maternal factors and breast milk composition. These include the lack of standard milk expression protocols, no specific time (time of day, foremilk or hindmilk) for expressing milk samples , and exclusive breastfeeding or the lack of information on the analysis of milk composition. In addition, most of the existing studies were conducted in the 1980s and 1990s and did not use separate up-to-date analyzers for protein, fat and lactose for milk composition analysis. Bzikowska-Jura et al., (2018) investigated the relationship between maternal nutrition and breast milk composition. However, in this study, mothers used a mix of hand and manual milking methods and the time elapsed since the baby's last feeding, which is another factor that may affect the content of breast milk, was not specified. Due to all these methodological differences, the effect of maternal diet on breast milk composition has not been clarified. These limitations may affect the actual assessment of these relationships. In this context, our study seeks answers to the effect of maternal diet on breast milk composition.

ELIGIBILITY:
Inclusion Criteria:

* - The mother is primigravida
* The mother has given birth naturally
* The mother is only breastfeeding her baby
* The mother is over 19 years old
* The mother's body mass index is within normal values (18.5 to 24.9)

Exclusion Criteria:

* The mother wants to quit her job.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — It should be done with breastfeeding mothers after birth. Breast milk has been analyzed.
Enrollment: 31 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Energy of breast milk as measured by Miris® HMA™ analyzer | Postpartum 23rd day
  Breast milk samples collected from each mother (10 mL) were stored at -18 °C and later thawed by a Nutrition and Dietetics researcher at 0-4 °C within 24 hours in the Nutrition and Dietetics Department Laboratory. To ensure reliability, each milk sample was analyzed twice. The energy content of the mature breast milk-energy (kcal/100 mL)-was determined using the Miris® Human Milk Analyzer™ (Miris AB, Uppsala, Sweden). The analysis results were recorded in the Breast Milk Tracking Form. "Breast milk energy content (kcal/100 mL), measured using Miris® Human Milk Analyzer Unit of Measure.
Protein of breast milk as measured by Miris® HMA™ analyzer | Postpartum 23rd day
  Breast milk samples collected from each mother (10 mL) were stored at -18 °C and later thawed by a Nutrition and Dietetics researcher at 0-4 °C within 24 hours in the Nutrition and Dietetics Department Laboratory. To ensure reliability, each milk sample was analyzed twice. The Protein content of the mature breast milk-protein (g/100 mL)-was determined using the Miris® Human Milk Analyzer™ (Miris AB, Uppsala, Sweden). The analysis results were recorded in the Breast Milk Tracking Form. "Breast milk protein content (g/100 mL), measured using Miris® Human Milk Analyzer Unit of Measure.
Fat of breast milk as measured by Miris® HMA™ analyzer | Postpartum 23rd day
  Breast milk samples collected from each mother (10 mL) were stored at -18 °C and later thawed by a Nutrition and Dietetics researcher at 0-4 °C within 24 hours in the Nutrition and Dietetics Department Laboratory. To ensure reliability, each milk sample was analyzed twice. The fat content of the mature breast milk-fat (g/100 mL)-was determined using the Miris® Human Milk Analyzer™ (Miris AB, Uppsala, Sweden). The analysis results were recorded in the Breast Milk Tracking Form. "Breast milk fat content (g/100 mL), measured using Miris® Human Milk Analyzer Unit of Measure.
Carbohydrate of breast milk as measured by Miris® HMA™ analyzer | Postpartum 23rd day
  Breast milk samples collected from each mother (10 mL) were stored at -18 °C and later thawed by a Nutrition and Dietetics researcher at 0-4 °C within 24 hours in the Nutrition and Dietetics Department Laboratory. To ensure reliability, each milk sample was analyzed twice. The Carbohydrate content of the mature breast milk-Carbohydrate (g/100 mL)-was determined using the Miris® Human Milk Analyzer™ (Miris AB, Uppsala, Sweden). The analysis results were recorded in the Breast Milk Tracking Form. "Breast milk Carbohydrate content (g/100 mL), measured using Miris® Human Milk Analyzer Unit of Measure.
Daily maternal energy intake (kcal/day), calculated using BeBiS 8.0 | postpartum days 20, 21, and 22
  Maternal food intake was assessed using the 24-Hour Food Consumption Record form. Data were analyzed using the Nutrition Information System (BeBiS 8.0), a software program adapted to Turkish dietary habits. Energy intake was calculated in kilocalories and reported as average daily intake.
  Protein: grams/100 mL
  Energy: kcal/100 mL
  24-Hour Dietary Recall Form
Daily maternal protein intake (gram/day), calculated using BeBiS 8.0 | postpartum days 20, 21, and 22
  Maternal food intake was assessed using the 24-Hour Food Consumption Record form. Data were analyzed using the Nutrition Information System (BeBiS 8.0), a software program adapted to Turkish dietary habits.
  Protein: grams/100 mL
  24-Hour Dietary Recall Form
Daily maternal fat intake (gram/day), calculated using BeBiS 8.0 | postpartum days 20, 21, and 22
  Maternal food intake was assessed using the 24-Hour Food Consumption Record form. Data were analyzed using the Nutrition Information System (BeBiS 8.0), a software program adapted to Turkish dietary habits.
  Fat: grams/100 mL
  24-Hour Dietary Recall Form
Daily maternal Carbohydrate intake (gram/day), calculated using BeBiS 8.0 | postpartum days 20, 21, and 22
  Maternal food intake was assessed using the 24-Hour Food Consumption Record form. Data were analyzed using the Nutrition Information System (BeBiS 8.0), a software program adapted to Turkish dietary habits.
  Carbohydrate : grams/100 mL
  24-Hour Dietary Recall Form

SECONDARY OUTCOMES:
The correlation between maternal dietary intake protein and protein content of breast milk | Between matched maternal-milk pairs after the 23rd day postpartum
  The correlation between maternal dietary intake protein, and protein content of breast milk will be assessed using Pearson correlation analysis. Each dietary variable will be compared to its respective breast milk component.
The correlation between maternal dietary intake energy and energy content of breast milk | Between matched maternal-milk pairs after the 23rd day postpartum
  The correlation between maternal dietary intake energy, and energy content of breast milk will be assessed using Pearson correlation analysis. Each dietary variable will be compared to its respective breast milk component.
The correlation between maternal dietary intake fat and fat content of breast milk | Between matched maternal-milk pairs after the 23rd day postpartum
  The correlation between maternal dietary intake fat and fat content of breast milk will be assessed using Pearson correlation analysis. Each dietary variable will be compared to its respective breast milk component.
The correlation between maternal dietary intake Carbohydrate and Carbohydrate content of breast milk | Between matched maternal-milk pairs after the 23rd day postpartum
  The correlation between maternal dietary intake Carbohydrate and Carbohydrate content of breast milk will be assessed using Pearson correlation analysis. Each dietary variable will be compared to its respective breast milk component.

CONTACTS AND LOCATIONS:
Overall Officials: Hülya Karataş, Professor, Study Director — Harran University
Locations (1):
- Harran University, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE STUDY MAY BE PUBLISHED AFTER IT IS PUBLISHED